CLINICAL TRIAL: NCT05483998
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of TLC-2716 in Healthy Subjects
Brief Title: A Study to Evaluate Single and Multiple Doses of TLC-2716 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OrsoBio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2716-CL-101
Record Dates: First submitted 2022-07-27; First posted 2022-08-02 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Open to Sponsor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A: Single Ascending Dose (SAD) (Experimental): Part A will be comprised of up to 50 participants over 5 cohorts of 10. Each participant will receive a single oral dose of TLC-2716 or placebo at different dose levels (1 cohort per dose level).
  Interventions: Drug: TLC-2716; Other: Placebo
- Part B: Multiple Ascending Dose (MAD) (Experimental): Part B will be comprised of up to 50 healthy participants over 5 cohorts of 10. Each participant will receive 14 oral doses of TLC-2716 or placebo over 14 days (given once daily) at different dose levels (1 cohort per dose level).
  Interventions: Drug: TLC-2716; Other: Placebo
- Part C: Adaptive SAD and/or MAD (Experimental): Part C is an adaptive style where the dosing level is a single- or multiple-ascending dose design. Based on safety and pharmacokinetic data from Parts A and B, doses for Part C will be chosen. Part C will be comprised of up to 50 participants over 5 cohorts of 10. Each participant will receive an oral dose of TLC-2716 or placebo at different dose levels (1 cohort per dose level).
  Interventions: Drug: TLC-2716; Other: Placebo

INTERVENTIONS:
Drug: TLC-2716 — TLC-2716
Other: Placebo — Placebo to match

SUMMARY:
This phase 1 study is designed to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of TLC-2716 after single- and multiple-ascending doses in healthy subjects.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, sponsor-unblinded, and comprised of three parts: Part A (single-ascending dose), Part B (multiple-ascending dose), and Part C (adaptive single- and/or multiple-ascending dose).

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, healthy male or female subject between 18 and 55 years of age, inclusive
* Body mass index from 19 to 35 kg/m2, inclusive
* Estimated glomerular filtration rate ≥ 80 mL/min
* Normal liver biochemistry tests
* Screening laboratory evaluations (hematology, chemistry, and urinalysis) must fall within the normal range of the local laboratory's reference ranges unless the results have been determined by the investigator to have no clinical significance
* Subject must have either a normal 12-lead electrocardiogram (ECG) or one with abnormalities that are considered clinically insignificant by the investigator
* Females of childbearing potential must have a negative pregnancy test at Screening and clinic admission
* Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception
* Must, in the opinion of the investigator, be in good health based upon medical history and physical examination, including vital signs

Exclusion Criteria:

* Pregnant or lactating subjects
* Subjects with triglycerides ≥ 500 mg/dL
* Subjects with low-density lipoprotein ≥ 190 mg/dL
* Subjects who have any serious or active medical or psychiatric illness (including depression) that, in the opinion of the investigator, would interfere with the subject's treatment, assessment, or compliance with the protocol
* Subjects who have received any investigational compound within 30 days or 5 half-lives, whichever is longer, prior to study drug dosing
* Current alcohol abuse that is judged by the investigator to potentially interfere with the subject's compliance or safety
* Current substance abuse that is judged by the investigator to potentially interfere with the subject's compliance or safety
* A positive test result for human immunodeficiency virus (HIV-1) antibody, hepatitis B (HBV) surface antigen, or hepatitis C (HCV) antibody
* Subjects who have taken any prescription medications or over-the-counter medications, including herbal products, within 28 days prior to start of study drug dosing, with the exception of vitamins, acetaminophen (paracetamol), ibuprofen, and/or hormonal contraceptive medications
* Subjects who have been treated with systemic steroids, immunosuppressant therapies, or chemotherapeutic agents within 3 months prior to Screening or expected to receive these agents during the study (e.g., corticosteroids, immunoglobulins, and other immune- or cytokine-based therapies)
* Medical history of serious skin disease in the opinion of the investigator, such as but not limited to rash, food allergy, eczema, psoriasis, or urticaria
* Medical history of drug sensitivity or drug allergy (such as anaphylaxis or hepatoxicity)
* Presence or history of cardiovascular disease, including significant cardiovascular disease (including a history of myocardial infarction based on ECG and/or clinical history), history of cardiac conduction abnormalities (including any history of ventricular tachycardia), congestive heart failure, cardiomyopathy with left ventricular ejection fraction < 40%, a family history of Long QT Syndrome, or unexplained death in an otherwise healthy individual between the ages of 1 and 30 years
* Syncope, palpitations, or unexplained dizziness
* Implanted defibrillator or pacemaker
* Medical history of liver disease, including but not limited to alcoholic liver disease, autoimmune disorders (e.g., primary biliary cholangitis, primary sclerosing cholangitis, autoimmune hepatitis), drug-induced hepatotoxicity, Wilson disease, clinically significant iron overload, or alpha-1-antitrypsin deficiency)
* Severe peptic ulcer disease, gastroesophageal reflux disease, or other gastric acid hypersecretory conditions
* History of medical or surgical treatment that permanently alters intestinal absorption (e.g., gastric or intestinal surgery)
* Subjects who have received vaccination for COVID-19 within 14 days of Admission

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-06-18 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (TEAEs) in single ascending dose (SAD) compared to placebo | Up to Day 15
  TEAEs are AEs that occur following the start of treatment or AEs increasing in severity during treatment.
Number of subjects with clinically significant change from Baseline in vital signs in SAD | Day 1-Day 4, and Follow-up (after 11 days)
  Vital signs include blood pressure, heart rate, respiratory rate, and temperature.
Number of subjects with laboratory abnormalities in SAD | Up to 15 days
  Hematology and serum chemistry.
Number of subjects with electrocardiogram (ECG) abnormalities in SAD | Up to 15 days
  12-lead ECG.
Number of subjects with TEAEs in multiple ascending dose (MAD) compared to placebo | Up to Day 28
  TEAEs are AEs that occur following the start of treatment or AEs increasing in severity during treatment.
Number of subjects with clinically significant change from Baseline in vital signs in MAD | Day 1 - Day 3, Day 5, Day 7, Day 10, Day 14, Day 17, and Follow-up (after 11 days)
  Vital signs include blood pressure, heart rate, respiratory rate, and temperature.
Number of subjects with laboratory abnormalities in MAD | Up to 28 days
  Hematology and serum chemistry.
Number of subjects with ECG abnormalities in MAD | Up to 28 days
  12-lead ECG

SECONDARY OUTCOMES:
Plasma concentration of each dose of study drug to determine AUClast in SAD | Day 1: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 12, 24, 48, and 72 hours post-dose
  AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Plasma concentration of each dose of study drug to determine AUCinf in SAD | Day 1: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 12, 24, 48, and 72 hours post-dose
  AUCinf is defined as the concentration of drug extrapolated to infinite time.
Plasma concentration of each dose of study drug to determine %AUCexp in SAD | Day 1: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 12, 24, 48, and 72 hours post-dose
  %AUCexp is defined as the percentage of AUC extrapolated between AUClast and AUCinf.
Plasma concentration of each dose of study drug to determine CL/F in SAD | Day 1: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 12, 24, 48, and 72 hours post-dose
  CL/F is defined as the apparent oral clearance following administration of the drug.
Plasma concentration of each dose of study drug to determine Cmax in SAD | Day 1: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 12, 24, 48, and 72 hours post-dose
  Cmax is defined as the maximum concentration of drug.
Plasma concentration of each dose of study drug to determine Tmax in SAD | Day 1: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 12, 24, 48, and 72 hours post-dose
  Tmax is defined as the time (observed time point) of Cmax.
Plasma concentration of each dose of study drug to determine Clast in SAD | Day 1: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 12, 24, 48, and 72 hours post-dose
  Clast is defined as the last observable concentration of drug.
Plasma concentration of each dose of study drug to determine Tlast in SAD | Day 1: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 12, 24, 48, and 72 hours post-dose
  Tlast is defined as the time (observed time point) of Clast.
Plasma concentration of each dose of study drug to determine t1/2 in SAD | Day 1: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 12, 24, 48, and 72 hours post-dose
  t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Plasma concentration of each dose of study drug to determine λz in SAD | Day 1: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 12, 24, 48, and 72 hours post-dose
  λz is defined as the terminal elimination rate constant, estimated by linear regression of the terminal elimination phase of the log plasma concentration of drug versus time curve of the drug.
Plasma concentration of each dose of study drug to determine AUClast in MAD | Day 1, Day 3, Day 7, Day 14
  AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Plasma concentration of each dose of study drug to determine AUCtau in MAD | Day 1, Day 3, Day 7, Day 14
  AUCtau is the concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval).
Plasma concentration of each dose of study drug to determine Ctau in MAD | Day 1, Day 3, Day 7, Day 14
  Ctau is defined as the observed drug concentration at the end of the dosing interval.
Plasma concentration of each dose of study drug to determine CLss/F in MAD | Day 1, Day 3, Day 7, Day 14
  CLss/F is the total body clearance for extravascular administration divided by the fraction of dose absorbed.
Plasma concentration of each dose of study drug to determine Cmax in MAD | Day 1, Day 3, Day 7, Day 14
  Cmax is defined as the maximum concentration of drug.
Plasma concentration of each dose of study drug to determine Tmax in MAD | Day 1, Day 3, Day 7, Day 14
  Tmax is defined as the time (observed time point) of Cmax.
Plasma concentration of each dose of study drug to determine Clast in MAD | Day 1, Day 3, Day 7, Day 14
  Clast is defined as the last observable concentration of drug.
Plasma concentration of each dose of study drug to determine Tlast in MAD | Day 1, Day 3, Day 7, Day 14
  Tlast is defined as the time (observed time point) of Clast.
Plasma concentration of each dose of study drug to determine t1/2 in MAD | Day 1, Day 3, Day 7, Day 14
  t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Plasma concentration of each dose of study drug to determine λz in MAD | Day 1, Day 3, Day 7, Day 14
  λz is defined as the terminal elimination rate constant, estimated by linear regression of the terminal elimination phase of the log plasma concentration of drug versus time curve of the drug.

CONTACTS AND LOCATIONS:
Overall Officials: OrsoBio Study Director, Study Director — OrsoBio, Inc
Locations (1):
- OrsoBio Research Site, Auckland, New Zealand

REFERENCES:
- [Derived] Li X, Benegiamo G, Vijayakumar A, Sroda N, Kimura M, Huss RS, Weng S, Murakami E, Kirby BJ, von Alvensleben GVG, Kremoser C, Gane EJ, Takebe T, Myers RP, Subramanian GM, Auwerx J. An oral, liver-restricted LXR inverse agonist for dyslipidemia: preclinical development and phase 1 trial. Nat Med. 2026 Jan 16. doi: 10.1038/s41591-025-04169-6. Online ahead of print. PMID 41545590